CLINICAL TRIAL: NCT03389620
Title: Comparison of Cervical Transforaminal Epidural Corticosteroid Injections With Lateralized Interlaminar Epidural Corticosteroid Injections for Treatment of Cervicogenic Upper Extremity Radiculopathy
Brief Title: Transforaminal Versus Lateralized Interlaminar Cervical Epidurals
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00083262
Record Dates: First submitted 2017-12-26; First posted 2018-01-03 (Actual); Results first posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Cervicogenic Upper Extremity Radiculopathy
Keywords: CT-fluoroscopy; Corticosteroid injection
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transforaminal Cervical Epidural Corticosteroid Injections (Active Comparator)
  Interventions: Drug: dexamethasone
- Lateralized Interlaminar Epidural Corticosteroid Injections (Experimental)
  Interventions: Drug: dexamethasone

INTERVENTIONS:
Drug: dexamethasone — 0.8 mL of dexamethasone (10 mg/mL) will slowly be injected over a period of approximately 30 seconds

SUMMARY:
The purpose of this study is to compare two methods of giving epidural steroid injections for nerve pain in the arm that comes from the neck. An epidural steroid injection can be given in two different ways, either in the back of the spine within the neck or in the neck next to the nerve root going to the arm. Both are standard medical treatments. The investigators would like to see how effective these treatments are, and if there are any differences in effectiveness or safety between these two routes.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral cervicogenic upper extremity radiculopathy (with or without accompanying neck pain)
* Baseline numerical pain scale (NRS) score > 4

Exclusion Criteria:

* Recent (i.e., < 2 months) cervical spine surgery
* Recent (i.e., < 1 month) cervical epidural or upper extremity corticosteroid injection
* Contraindication or inability to the undergo procedure
* Inability to provide informed consent
* Expected inability to complete follow-up assessment
* Contraindication to receiving contrast material (precluding an epidurogram)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2023-07-16 (Actual); Study Completion 2023-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Amrhein, MD, Principal Investigator — Duke University
Locations (1):
- Duke Radiology and Orthopaedic Clinic, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with unilateral cervicogenic radiculopathy referred for a cervical epidural steroid injection were recruited from the outpatient Duke Radiology Spine Intervention Clinic.
Pre-assignment Details: This is not a crossover study.
Period: Overall Study
Arm/Group | Transforaminal Cervical Epidural Corticosteroid Injections | Lateralized Interlaminar Epidural Corticosteroid Injections
Started | 37 | 37
Completed | 32 | 36
Not Completed | 5 | 1
Not completed — Lost to Follow-up | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transforaminal Cervical Epidural Corticosteroid Injections | Lateralized Interlaminar Epidural Corticosteroid Injections | Total
Number analyzed (Participants) | 37 | 37 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.68 (14.11) | 54.49 (11.94) | 55.58 (13.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 21 | 43
  Male | 15 | 16 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 35 | 36 | 71
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 9 | 8 | 17
  White | 25 | 29 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37 | 37 | 74

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Numerical Rating Scale (Averaged Over Past 24 Hours)
Description: The pain numerical rating scale (NRS) is a well-validated tool for quantitatively assessing patients' pain. The NRS asks patients to rate their current pain intensity on an 11-point scale ranging from 0 ("no pain") to 10 ("worst possible pain")
Time Frame: Baseline to 2 months
Population: Data not collected on 3 Transforaminal Cervical Epidural Corticosteroid Injection participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transforaminal Cervical Epidural Corticosteroid Injections | Lateralized Interlaminar Epidural Corticosteroid Injections
Number analyzed (Participants) | 34 | 37
score on a scale | -3.38 (2.50) | -2.30 (2.20)
Statistical Analysis 1: Comparison: Transforaminal Cervical Epidural Corticosteroid Injections vs Lateralized Interlaminar Epidural Corticosteroid Injections; Test type: Non-Inferiority — Based on previous literature indicating that the minimum clinical threshold for change in NRS pain score is 2 points, a non-inferiority margin of differential change between treatment arms of 2 points at the 2 month time point following the surgical procedure was specified, assuming the true difference between treatment arms is zero; p = 0.057, t-test, 1 sided

2. Secondary Outcome: Change in Pain Numerical Rating Scale (Averaged Over Past 24 Hours)
Description: as for outcome 1
Time Frame: Baseline, 2 weeks, 4 months
Population: Participants with data collected at each timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transforaminal Cervical Epidural Corticosteroid Injections | Lateralized Interlaminar Epidural Corticosteroid Injections
Number analyzed (Participants) | 37 | 37
score on a scale
  Baseline to 2 weeks | -2.51 (2.58) | -3.03 (2.37)
  Baseline to 4 months: number analyzed (Participants) | 32 | 36
  Baseline to 4 months | -3.44 (3.15) | -3.31 (2.40)
Statistical Analysis 1: Comparison: Transforaminal Cervical Epidural Corticosteroid Injections vs Lateralized Interlaminar Epidural Corticosteroid Injections; Baseline to 2 weeks; Test type: Superiority; p = 0.376, t-test, 2 sided
Statistical Analysis 2: Comparison: Transforaminal Cervical Epidural Corticosteroid Injections vs Lateralized Interlaminar Epidural Corticosteroid Injections; Baseline to 4 months; Test type: Superiority; p = 0.848, t-test, 2 sided

3. Secondary Outcome: Change in Neck Disability Index (NDI)
Description: The NDI a well-validated measurement tool that contains 10 items: seven related to activities of daily living, two related to pain, and one related to concentration. Each item is scored from 0 to 5 and the total score is expressed as a percentage, with higher scores corresponding to greater disability.
Time Frame: Baseline, 2 weeks, 2 months, 4 months
Population: Participants with data collected at each timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transforaminal Cervical Epidural Corticosteroid Injections | Lateralized Interlaminar Epidural Corticosteroid Injections
Number analyzed (Participants) | 37 | 37
score on a scale
  Baseline to 2 weeks | -10.97 (15.62) | -9.30 (12.58)
  Baseline to 2 months: number analyzed (Participants) | 34 | 37
  Baseline to 2 months | -10.24 (16.03) | -8.00 (16.51)
  Baseline to 4 months: number analyzed (Participants) | 32 | 36
  Baseline to 4 months | -14.25 (22.04) | -14.00 (16.18)
Statistical Analysis 1: Comparison: Transforaminal Cervical Epidural Corticosteroid Injections vs Lateralized Interlaminar Epidural Corticosteroid Injections; Baseline to 2 weeks; Test type: Superiority; p = 0.613, t-test, 2 sided
Statistical Analysis 2: Comparison: Transforaminal Cervical Epidural Corticosteroid Injections vs Lateralized Interlaminar Epidural Corticosteroid Injections; Baseline to 2 months; Test type: Superiority; p = 0.565, t-test, 2 sided
Statistical Analysis 3: Comparison: Transforaminal Cervical Epidural Corticosteroid Injections vs Lateralized Interlaminar Epidural Corticosteroid Injections; Baseline to 4 months; Test type: Superiority; p = 0.958, t-test, 2 sided

4. Secondary Outcome: Change in EuroQol-5 Dimension (EQ-5D) Visual Analog Scale (VAS)
Description: EQ-5D is a standardized measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal. It is a well-validated tool for health status measurement, and for health quality-of-life in cervicogenic radicular pain. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labeled 'The best health you can imagine' (100) and 'The worst health you can imagine' (0).
Time Frame: Baseline, 2 weeks, 2 months, 4 months
Population: Participants with data collected at each timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transforaminal Cervical Epidural Corticosteroid Injections | Lateralized Interlaminar Epidural Corticosteroid Injections
Number analyzed (Participants) | 37 | 37
score on a scale
  Baseline to 2 weeks | 5.49 (25.40) | -0.38 (21.51)
  Baseline to 2 months: number analyzed (Participants) | 34 | 37
  Baseline to 2 months | 3.79 (23.58) | -1.03 (20.69)
  Baseline to 4 months: number analyzed (Participants) | 32 | 36
  Baseline to 4 months | 1.48 (37.45) | 2.69 (18.15)
Statistical Analysis 1: Comparison: Transforaminal Cervical Epidural Corticosteroid Injections vs Lateralized Interlaminar Epidural Corticosteroid Injections; Baseline to 2 weeks; Test type: Superiority; p = 0.287, t-test, 2 sided
Statistical Analysis 2: Comparison: Transforaminal Cervical Epidural Corticosteroid Injections vs Lateralized Interlaminar Epidural Corticosteroid Injections; Baseline to 2 months; Test type: Superiority; p = 0.365, t-test, 2 sided
Statistical Analysis 3: Comparison: Transforaminal Cervical Epidural Corticosteroid Injections vs Lateralized Interlaminar Epidural Corticosteroid Injections; Baseline to 4 months; Test type: Superiority; p = 0.867, t-test, 2 sided

5. Secondary Outcome: Change in EuroQol-5 Dimension (EQ-5D) Index Score
Description: EQ-5D is a standardized measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal. It is a well-validated tool for health status measurement, and for health quality-of-life in cervicogenic radicular pain. The index score was derived using the time trade-off (TTO) valuation method and ranges from approximately 0 (dead) to 1 (full health), with negative values indicating health states worse than death.
Time Frame: Baseline, 2 weeks, 2 months, 4 months
Population: Participants with data collected at each timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transforaminal Cervical Epidural Corticosteroid Injections | Lateralized Interlaminar Epidural Corticosteroid Injections
Number analyzed (Participants) | 37 | 37
score on a scale
  Baseline to 2 weeks | 0.085 (0.238) | 0.137 (0.202)
  Baseline to 2 months: number analyzed (Participants) | 34 | 37
  Baseline to 2 months | 0.088 (0.205) | 0.131 (0.205)
  Baseline to 4 months: number analyzed (Participants) | 32 | 36
  Baseline to 4 months | 0.145 (0.257) | 0.172 (0.259)
Statistical Analysis 1: Comparison: Transforaminal Cervical Epidural Corticosteroid Injections vs Lateralized Interlaminar Epidural Corticosteroid Injections; Baseline to 2 weeks; Test type: Superiority; p = 0.311, t-test, 2 sided
Statistical Analysis 2: Comparison: Transforaminal Cervical Epidural Corticosteroid Injections vs Lateralized Interlaminar Epidural Corticosteroid Injections; Baseline to 2 months; Test type: Superiority; p = 0.377, t-test, 2 sided
Statistical Analysis 3: Comparison: Transforaminal Cervical Epidural Corticosteroid Injections vs Lateralized Interlaminar Epidural Corticosteroid Injections; Baseline to 4 months; Test type: Superiority; p = 0.668, t-test, 2 sided

6. Secondary Outcome: Change in Work Ability Index (WAI) Absenteeism
Description: The Work Ability Index (WAI) is a validated, reliable measure of a worker's ability to do his or her job that has been shown to predict work disability, retirement and mortality. The WAI is scored on a scale of 7 to 49, where higher scores indicate better work ability.
Time Frame: Baseline, 2 weeks, 2 months, 4 months
Population: Employed participants with data collected at each timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transforaminal Cervical Epidural Corticosteroid Injections | Lateralized Interlaminar Epidural Corticosteroid Injections
Number analyzed (Participants) | 20 | 22
score on a scale
  Baseline to 2 weeks | -11.76 (31.82) | -8.81 (35.85)
  Baseline to 2 months: number analyzed (Participants) | 16 | 21
  Baseline to 2 months | -13.66 (30.09) | -11.40 (38.96)
  Baseline to 4 months: number analyzed (Participants) | 16 | 19
  Baseline to 4 months | -9.09 (25.09) | -12.37 (27.28)
Statistical Analysis 1: Comparison: Transforaminal Cervical Epidural Corticosteroid Injections vs Lateralized Interlaminar Epidural Corticosteroid Injections; Baseline to 2 weeks; Test type: Superiority; p = 0.794, t-test, 2 sided
Statistical Analysis 2: Comparison: Transforaminal Cervical Epidural Corticosteroid Injections vs Lateralized Interlaminar Epidural Corticosteroid Injections; Baseline to 2 months; Test type: Superiority; p = 0.843, t-test, 2 sided
Statistical Analysis 3: Comparison: Transforaminal Cervical Epidural Corticosteroid Injections vs Lateralized Interlaminar Epidural Corticosteroid Injections; Baseline to 4 months; Test type: Superiority; p = 0.713, t-test, 2 sided

7. Secondary Outcome: Change in Work Ability Index (WAI) Presenteeism
Description: as for outcome 6
Time Frame: Baseline, 2 weeks, 2 months, 4 months
Population: Employed participants with data collected at each timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transforaminal Cervical Epidural Corticosteroid Injections | Lateralized Interlaminar Epidural Corticosteroid Injections
Number analyzed (Participants) | 21 | 22
score on a scale
  Baseline to 2 weeks | -8.95 (21.58) | -19.55 (27.68)
  Baseline to 2 months: number analyzed (Participants) | 19 | 22
  Baseline to 2 months | -8.95 (22.58) | -19.09 (40.93)
  Baseline to 4 months: number analyzed (Participants) | 17 | 20
  Baseline to 4 months | -26.50 (43.44) | -18.82 (24.46)
Statistical Analysis 1: Comparison: Transforaminal Cervical Epidural Corticosteroid Injections vs Lateralized Interlaminar Epidural Corticosteroid Injections; Baseline to 2 weeks; Test type: Superiority; p = 0.177, t-test, 2 sided
Statistical Analysis 2: Comparison: Transforaminal Cervical Epidural Corticosteroid Injections vs Lateralized Interlaminar Epidural Corticosteroid Injections; Baseline to 2 months; Test type: Superiority; p = 0.325, t-test, 2 sided
Statistical Analysis 3: Comparison: Transforaminal Cervical Epidural Corticosteroid Injections vs Lateralized Interlaminar Epidural Corticosteroid Injections; Baseline to 4 months; Test type: Superiority; p = 0.505, t-test, 2 sided

8. Secondary Outcome: Change in Work Ability Index (WAI) Work Productivity Loss
Description: as for outcome 6
Time Frame: Baseline, 2 weeks, 2 months, 4 months
Population: Employed participants with data collected at each timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transforaminal Cervical Epidural Corticosteroid Injections | Lateralized Interlaminar Epidural Corticosteroid Injections
Number analyzed (Participants) | 20 | 22
score on a scale
  Baseline to 2 weeks | -18.97 (18.80) | -20.79 (34.32)
  Baseline to 2 months: number analyzed (Participants) | 19 | 22
  Baseline to 2 months | -8.95 (22.58) | -19.09 (40.93)
  Baseline to 4 months: number analyzed (Participants) | 16 | 19
  Baseline to 4 months | -21.16 (25.84) | -26.37 (45.47)
Statistical Analysis 1: Comparison: Transforaminal Cervical Epidural Corticosteroid Injections vs Lateralized Interlaminar Epidural Corticosteroid Injections; Baseline to 2 weeks; Test type: Superiority; p = 0.811, t-test, 2 sided
Statistical Analysis 2: Comparison: Transforaminal Cervical Epidural Corticosteroid Injections vs Lateralized Interlaminar Epidural Corticosteroid Injections; Baseline to 2 months; Test type: Superiority; p = 0.325, t-test, 2 sided
Statistical Analysis 3: Comparison: Transforaminal Cervical Epidural Corticosteroid Injections vs Lateralized Interlaminar Epidural Corticosteroid Injections; Baseline to 4 months; Test type: Superiority; p = 0.674, t-test, 2 sided

9. Secondary Outcome: Change in Work Ability Index (WAI) Activity Impairment
Description: as for outcome 6
Time Frame: Baseline, 2 weeks, 2 months, 4 months
Population: Employed participants with data collected at each timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transforaminal Cervical Epidural Corticosteroid Injections | Lateralized Interlaminar Epidural Corticosteroid Injections
Number analyzed (Participants) | 20 | 22
score on a scale
  Baseline to 2 weeks | -13.51 (31.20) | -12.70 (25.35)
  Baseline to 2 months: number analyzed (Participants) | 19 | 22
  Baseline to 2 months | -9.12 (32.13) | -14.32 (32.54)
  Baseline to 4 months: number analyzed (Participants) | 16 | 20
  Baseline to 4 months | -18.18 (32.74) | -21.11 (33.87)
Statistical Analysis 1: Comparison: Transforaminal Cervical Epidural Corticosteroid Injections vs Lateralized Interlaminar Epidural Corticosteroid Injections; Baseline to 2 weeks; Test type: Superiority; p = 0.903, t-test, 2 sided
Statistical Analysis 2: Comparison: Transforaminal Cervical Epidural Corticosteroid Injections vs Lateralized Interlaminar Epidural Corticosteroid Injections; Baseline to 2 months; Test type: Superiority; p = 0.500, t-test, 2 sided
Statistical Analysis 3: Comparison: Transforaminal Cervical Epidural Corticosteroid Injections vs Lateralized Interlaminar Epidural Corticosteroid Injections; Baseline to 4 months; Test type: Superiority; p = 0.716, t-test, 2 sided

10. Secondary Outcome: Number of Participants With Minor Adverse Events
Time Frame: Immediately post-procedure, 2 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Transforaminal Cervical Epidural Corticosteroid Injections | Lateralized Interlaminar Epidural Corticosteroid Injections
Number analyzed (Participants) | 37 | 37
Participants
  Immediately post-procedure | 3 | 6
  2 days post procedure | 4 | 5
Statistical Analysis 1: Comparison: Transforaminal Cervical Epidural Corticosteroid Injections vs Lateralized Interlaminar Epidural Corticosteroid Injections; Immediately post-procedure; Test type: Superiority; p = 0.461, Fisher Exact
Statistical Analysis 2: Comparison: Transforaminal Cervical Epidural Corticosteroid Injections vs Lateralized Interlaminar Epidural Corticosteroid Injections; 2 days post procedure; Test type: Superiority; p = 1.00, Fisher Exact

11. Secondary Outcome: Number of Participants With Major Adverse Events
Time Frame: Immediately post-procedure, 2 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Transforaminal Cervical Epidural Corticosteroid Injections | Lateralized Interlaminar Epidural Corticosteroid Injections
Number analyzed (Participants) | 37 | 37
Participants
  Immediately post-procedure | 0 | 0
  2 days post procedure | 0 | 0

12. Other Pre Specified Outcome: Number of Participants With Inadvertent Intravascular Contrast Injections
Time Frame: During procedure
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Number of Participants With Contrast Spread Into the Medial Half of the Neuroforamen
Time Frame: During procedure
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 2 days post-procedure
Arm/Group | Transforaminal Cervical Epidural Corticosteroid Injections | Lateralized Interlaminar Epidural Corticosteroid Injections
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/37
Other Adverse Events (participants affected / at risk) | 6/37 | 8/37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Transforaminal Cervical Epidural Corticosteroid Injections (N=37) | Lateralized Interlaminar Epidural Corticosteroid Injections (N=37)
Nausea (Gastrointestinal disorders) | 1 | 2
Headache (General disorders) | 3 | 4
Vasovagal (General disorders) | 0 | 2
Lightheadedness (General disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-15): https://cdn.clinicaltrials.gov/large-docs/20/NCT03389620/Prot_SAP_000.pdf